CLINICAL TRIAL: NCT02714699
Title: Randomized Clinical Trial of Oral Hyoscine Butyl Bromide Versus Diclofenac Potassium in Reducing Pain During Office Hysteroscopy
Brief Title: Oral Hyoscine Butyl Bromide Versus Diclofenac Potassium Before Office Hysteroscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HB-OH
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Endoscopy
MeSH Terms: interventions — Diclofenac; Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- diclofenac potassium (Experimental): oral diclofenac potassium
  Interventions: Drug: diclofenac potassium
- hyoscine butyl bromide (Active Comparator): oral hyoscine butyl bromide
  Interventions: Drug: hyoscine butyl bromide
- placebo (Placebo Comparator): oral placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: diclofenac potassium — patients will take oral diclofenac potassium; two tablets (cataflam 25 mg) and one tablet placebo one hour before the procedure
  Other Names: cataflam
  Arms: diclofenac potassium
Drug: hyoscine butyl bromide — patients will take oral hyoscine-N- butyl bromide; 2 tablets (buscopan 10 mg) one hour before the procedure
  Other Names: buscopan
  Arms: hyoscine butyl bromide
Drug: placebo — patients will take oral placebo; 2 tablets one hour before the procedure
  Arms: placebo

SUMMARY:
The study aims to determine the efficacy of oral hyoscine butyl bromide versus diclofenac potassium on the pain scores during office hysteroscopy

ELIGIBILITY:
Inclusion Criteria:

1. Patients that must perform a diagnostic hysteroscopy.
2. Acceptance to participate in the study.
3. Signed informed consent.
4. Not taking analgesics (acetaminophen, ibuprofen, mefenamic acid) before admission.
5. Absence of sedative use before admission

Exclusion Criteria:

1. Hypersensitivity to drugs
2. refusal of the patient
3. Patients are pregnant.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Mean pain score during hysteroscopy | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes